CLINICAL TRIAL: NCT01696929
Title: An Open-Label Trial of Tocilizumab in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brian Miller (Other)
Responsible Party: Sponsor-Investigator, Brian Miller, Assistant Professor, Augusta University
Organization: Augusta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000405
Record Dates: First submitted 2012-09-24; First posted 2012-10-02 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
Keywords: tocilizumab; safety; tolerability; efficacy; schizophrenia; improvement; cognition; psychotic symptoms; baseline IL-6 levels
MeSH Terms: conditions — Schizophrenia | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tocilizumab (Experimental): Following a screening evaluation, participants will receive two infusions of tocilizumab, one at baseline and another at week 4 of the study. All subjects will receive a 4 mg/kg infusion of tocilizumab, the recommended starting dose for adults with rheumatoid arthritis.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Therapeutic/Pharmacologic Class of Drug:
  Tocilizumab is a recombinant humanized anti-human interleukin-6 (IL-6) receptor monoclonal antibody of the immunoglobulin (Ig) gamma-1 subclass.
  Type of Dosage Form:
  Concentrate for solution for infusion.
  Route of Administration:
  Intravenous (i.v.) infusion.
  Other Names: Brand Name: Actemra; NDA/Serial Number: STN 125276/S022 (Cross ref: IND 11972)

SUMMARY:
This study is a Phase 1 clinical trail to determine the safety, tolerability, and efficacy of Tocilizumab (Actemra) as an adjunct to antipsychotic medications in stable outpatients with schizophrenia. Tocilizumab (structural formula C6428H9976N1720O2018S42) is a recombinant humanized anti-human interleukin-6 (IL-6) receptor monoclonal antibody of the immunoglobulin (Ig) gamma-1 subclass. Tocilizumab is formulated as a concentrate for solution for infusion, and will be administered by intravenous infusion.

The investigators propose an 8-week trial to determine the safety, tolerability, and effectiveness of tocilizumab, given in addition to antipsychotic medications, in 10 stable outpatients with schizophrenia. The investigators hypothesize that tocilizumab will be associated with clinically significant improvement in cognition and total psychotic symptoms over the course of the trial. Tocilizumab is administered as an intravenous infusion every 4 weeks. Following a screening evaluation, participants will receive two infusions of tocilizumab, one at baseline and another at week 4 of the study. The investigators will measure changes in cognitive function and symptoms over an 8-week period. Complementing previous positive clinical trials of non-steroidal anti-inflammatory drugs, this would be a "proof-of-concept" study that targeting specific cytokines is a viable treatment for schizophrenia.

Interleukin 6 and its receptor were discovered and cloned at Osaka University, Japan, by Tadamitsu Kishimoto in the 1980s. In 1997, Chugai Pharmaceuticals began the clinical development of tocilizumab for the treatment of rheumatoid arthritis. Clinical studies for Castleman's disease and systemic juvenile idiopathic arthritis started in 2001 and 2002, respectively. Hoffmann-La Roche co-developed the drug due to a license agreement in 2003.

Data presented in 2008 showed the effectiveness of tocilizumab in combination therapy with methotrexate for rheumatoid arthritis treatment. In further studies, it was effective and generally well tolerated when administered either as monotherapy or in combination with conventional disease-modifying antirheumatic drugs in adult patients with moderate to severe rheumatoid arthritis.

DETAILED DESCRIPTION:
Schizophrenia is a chronic, debilitating disorder with life-long consequences on affected individuals and families. Schizophrenia is also associated with impaired cognition or thinking, which persists despite currently available treatments, and is an important determinant of quality of life and overall function. Associations between immune system abnormalities and schizophrenia, in particular increased inflammation, are one of the more enduring findings in the field. Four of six trials found that treatment with non-steroidal anti-inflammatory drugs (NSAIDs) was associated with significant improvement in psychopathology (Muller et al., 2010a; Muller et al., 2010b). Serum cytokine levels predicted response in two studies (Laan et al., 2010; Muller et al., 2004), and another study found a trend for improved cognition (Muller et al., 2005) with adjunctive NSAID treatment. These findings provide important empirical support for a pathophysiological role for inflammation in a subset of patients with schizophrenia.

Cytokines are key regulators of inflammation that exert effects in the periphery and the brain. IL-6 is a cytokine produced by peripheral blood leukocytes, and central nervous system microglia and astrocytes. Serum IL-6 levels are increased in patients with schizophrenia, and two studies reported significant positive correlations between IL-6 and total psychopathology at baseline and following antipsychotic treatment (Miller et al., 2011). Schizophrenia is associated with impaired cognition, which persists despite current treatments, and is an important determinant of quality of life and overall function. In populations outside of schizophrenia, higher serum IL-6 levels are associated with poorer cognition, cognitive decline, and smaller hippocampal gray matter volume (Marsland et al., 2006; Marsland et al., 2008). In a first-episode psychosis sample, IL-6 messenger ribonucleic acid expression was a significant predictor of smaller left hippocampal volume (Mondelli et al., 2011).

Several other lines of evidence provide a theoretical background for targeting IL-6 in schizophrenia. Polymorphisms of the gene for IL-6 (Paul-Samojedny et al., 2010) and its receptor (Sun et al., 2008) have been associated with schizophrenia. In mice, a single maternal injection of IL-6 during pregnancy caused prepulse and latent inhibition deficits in the adult offspring (Smith et al., 2007). Prenatal maternal infections are a replicated risk factor for schizophrenia (Brown and Derkits, 2010). In a rat prenatal immune activation model, adult offspring have increased serum IL-6 levels, at an age with homology to the usual age of onset of schizophrenia, that are significantly decreased following treatment with haloperidol (Romero et al., 2007; Romero et al., 2010). Another animal study found that ketamine-induced neuronal production of IL-6 is responsible for the activation of brain NADPH-oxidase and subsequent dysfunction of fast-spiking parvalbumin-expressing interneurons (Behrens et al., 2008). These findings provide further support for a potential role of IL-6 in the pathophysiology of schizophrenia.

In our Preliminary Study, patients with schizophrenia, age 18-70 and taking non-clozapine antipsychotics, had a fasting blood draw for serum cytokines, and assessment of psychopathology, including cognition. Subjects were not taking NSAIDs, and had no history of immune disorders, illicit drug use in the past month, or antibiotic use in the past 2 weeks. In 39 patients, after controlling for potential confounding effects of age, sex, race, smoking, BMI, socioeconomic status, serum cortisol, psychotropic medications, intelligence quotient, and severity of psychopathology, higher serum IL-6 levels predicted greater cognitive impairment, measured by the Brief Assessment of Cognition in Schizophrenia (BACS) composite score, in a linear regression model (p=0.002, Figure 1). Higher IL-6 levels were also associated with significantly lower scores on the Verbal Memory (r=-0.40, p<0.01) and Motor Speed (r=-0.42, p<0.01) subtests of the BACS.

In the first year, one clinical trial is planned. We will conduct an 8-week open-label trial to determine the safety, tolerability, and efficacy of tocilizumab as an adjunct to antipsychotic medications in 10 stable outpatients with schizophrenia.

Tocilizumab has not been used before in the treatment of schizophrenia, and using it this way is experimental. The risks that have been found in people with rheumatoid arthritis are known, but there may be unknown risks when used in schizophrenia. Clinically significant adverse drug reactions include anaphylaxis (0.4%), infections (0.1-7.8%), intestinal perforation, neutropenia (7.0%), and cardiac failure. Known side effects of tocilizumab that are common include: increase in hepatic enzymes (AST, ALT), hypertension, headache, neutropenia, infusion-related reactions, upper respiratory tract infections, and nasopharyngitis.

Less common side effects include: peripheral edema, dizziness, rash, increased total cholesterol and LDL, hypothyroidism, diarrhea, abdominal pain, mouth ulcerations, gastric ulcer, stomatitis, weight gain, gastritis, thrombocytopenia, leukopenia, increased bilirubin, conjunctivitis, nephrolithiasis, bronchitis, cough, dyspnea, herpes simplex. Rare side effects include: cellulitis, fungal infections, diverticulitis, gastroenteritis, herpes zoster, hypertriglyceridemia, malignancy (including breast and colon), multiple sclerosis, otitis media, pneumonia, sepsis, tuberculosis, urinary tract infections, and varicella.

Subjects with schizophrenia will be accessed from outpatient psychiatry clinic at Georgia Health Sciences University or other satellite collaborative sites. The study has 5 visits: screening, baseline, and 2, 4, and 8 weeks. At Screening, all subjects will be administered the evaluation to sign consent, informed consent, and the structured clinical interview for Diagnostic and Statistical Manual psychosis and affective disorders modules. We will perform a medical history and physical exam, fasting labs (CBC, Complete Metabolic Panel, lipid panel, urinalysis, and urine drug screen (UDS)), a tuberculin skin test, and a 12-lead electrocardiogram. At Baseline, we will perform the Positive and Negative Syndrome Scale, BACS, and Clinical Global Impressions scale (CGI), and draw blood for IL-6 and high-sensitivity c-reactive protein (hsCRP). All subjects will receive a 4 mg/kg infusion of tocilizumab, the recommended starting dose for adults with rheumatoid arthritis. We will contact the subjects by phone on day 1 and 7 after the infusion to assess for any infusion-related events. At Week 2 and 4, we will perform an interval history, physical exam, Positive and Negative Syndrome Scale, BACS, and CGI. Different versions of the BACS will be used to avoid practice effects. At Week 4, we will obtain fasting labs (CBC, Complete Metabolic Panel, lipid panel, IL-6, hsCRP, and UDS), and subjects will receive a 4 mg/kg infusion of tocilizumab, We will contact the subjects by phone day 1 and 7 after the second infusion to assess for any infusion-related events. At Week 8, we will perform an interval history, physical exam, and administer the Positive and Negative Syndrome Scale, BACS, CGI, and obtain fasting labs (CBC, Complete Metabolic Panel, lipid panel, IL-6, hsCRP, and UDS). Patients will be withdrawn if they meet any exclusion criterion at any time point.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* age 18-50
* capable of giving informed consent
* diagnosis of schizophrenia
* stable based on clinical judgement, no psychiatric hospitalizations in past 3 months, and on the same psychotropic medications for >4 weeks
* taking a non-clozapine antipsychotic

Exclusion Criteria:

* imminent danger to self/others
* antibiotic use in the past 2 weeks
* current scheduled use of immunomodulatory agents
* history of an immune disorder
* illicit drug use in the past 30 days
* any unstable or untreated medical condition
* history of gastrointestinal ulcers, diverticulitis, malignancy, central nervous system demyelinating disorder, seizure disorder, or tuberculosis
* low absolute neutrophil (<2000) or platelet (<100,000) count
* abnormal hepatic (AST or ALT >1.5 times the upper limit of normal) or renal (BUN or creatinine>1.5 times the upper limit of normal) function
* any abnormal lab test result judged to be clinically significant
* active, chronic or recurrent infections
* pregnancy
* breastfeeding
* female and of child-bearing potential who is not using any contraception

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Miller, MD, PhD, MPH, Principal Investigator — Augusta University - Department of Psychiatry and Health Behavior
Locations (1):
- Georgia Health Sciences University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller N. COX-2 inhibitors as antidepressants and antipsychotics: clinical evidence. Curr Opin Investig Drugs. 2010 Jan;11(1):31-42. PMID 20047157
- [Background] Muller N, Krause D, Dehning S, Musil R, Schennach-Wolff R, Obermeier M, Moller HJ, Klauss V, Schwarz MJ, Riedel M. Celecoxib treatment in an early stage of schizophrenia: results of a randomized, double-blind, placebo-controlled trial of celecoxib augmentation of amisulpride treatment. Schizophr Res. 2010 Aug;121(1-3):118-24. doi: 10.1016/j.schres.2010.04.015. Epub 2010 May 31. PMID 20570110
- [Background] Muller N, Ulmschneider M, Scheppach C, Schwarz MJ, Ackenheil M, Moller HJ, Gruber R, Riedel M. COX-2 inhibition as a treatment approach in schizophrenia: immunological considerations and clinical effects of celecoxib add-on therapy. Eur Arch Psychiatry Clin Neurosci. 2004 Feb;254(1):14-22. doi: 10.1007/s00406-004-0478-1. PMID 14991374
- [Background] Laan W, Grobbee DE, Selten JP, Heijnen CJ, Kahn RS, Burger H. Adjuvant aspirin therapy reduces symptoms of schizophrenia spectrum disorders: results from a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2010 May;71(5):520-7. doi: 10.4088/JCP.09m05117yel. PMID 20492850
- [Background] Muller N, Riedel M, Schwarz MJ, Engel RR. Clinical effects of COX-2 inhibitors on cognition in schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2005 Apr;255(2):149-51. doi: 10.1007/s00406-004-0548-4. Epub 2004 Nov 19. PMID 15549344
- [Background] Miller BJ, Buckley P, Seabolt W, Mellor A, Kirkpatrick B. Meta-analysis of cytokine alterations in schizophrenia: clinical status and antipsychotic effects. Biol Psychiatry. 2011 Oct 1;70(7):663-71. doi: 10.1016/j.biopsych.2011.04.013. Epub 2011 Jun 8. PMID 21641581
- [Background] Marsland AL, Petersen KL, Sathanoori R, Muldoon MF, Neumann SA, Ryan C, Flory JD, Manuck SB. Interleukin-6 covaries inversely with cognitive performance among middle-aged community volunteers. Psychosom Med. 2006 Nov-Dec;68(6):895-903. doi: 10.1097/01.psy.0000238451.22174.92. PMID 17132839
- [Background] Marsland AL, Gianaros PJ, Abramowitch SM, Manuck SB, Hariri AR. Interleukin-6 covaries inversely with hippocampal grey matter volume in middle-aged adults. Biol Psychiatry. 2008 Sep 15;64(6):484-90. doi: 10.1016/j.biopsych.2008.04.016. Epub 2008 Jun 2. PMID 18514163
- [Background] Mondelli V, Cattaneo A, Murri MB, Di Forti M, Handley R, Hepgul N, Miorelli A, Navari S, Papadopoulos AS, Aitchison KJ, Morgan C, Murray RM, Dazzan P, Pariante CM. Stress and inflammation reduce brain-derived neurotrophic factor expression in first-episode psychosis: a pathway to smaller hippocampal volume. J Clin Psychiatry. 2011 Dec;72(12):1677-1684. doi: 10.4088/JCP.10m06745. Epub 2011 May 18. PMID 21672499
- [Background] Paul-Samojedny M, Kowalczyk M, Suchanek R, Owczarek A, Fila-Danilow A, Szczygiel A, Kowalski J. Functional polymorphism in the interleukin-6 and interleukin-10 genes in patients with paranoid schizophrenia--a case-control study. J Mol Neurosci. 2010 Sep;42(1):112-9. doi: 10.1007/s12031-010-9365-6. PMID 20393813
- [Background] Sun S, Wang F, Wei J, Cao LY, Qi LY, Xiu MH, Chen S, Li XH, Kosten TA, Kosten TR, Zhang XY. Association between interleukin-6 receptor polymorphism and patients with schizophrenia. Schizophr Res. 2008 Jul;102(1-3):346-7. doi: 10.1016/j.schres.2008.04.018. Epub 2008 May 27. No abstract available. PMID 18508242
- [Background] Smith SE, Li J, Garbett K, Mirnics K, Patterson PH. Maternal immune activation alters fetal brain development through interleukin-6. J Neurosci. 2007 Oct 3;27(40):10695-702. doi: 10.1523/JNEUROSCI.2178-07.2007. PMID 17913903
- [Background] Brown AS, Derkits EJ. Prenatal infection and schizophrenia: a review of epidemiologic and translational studies. Am J Psychiatry. 2010 Mar;167(3):261-80. doi: 10.1176/appi.ajp.2009.09030361. Epub 2010 Feb 1. PMID 20123911
- [Background] Romero E, Ali C, Molina-Holgado E, Castellano B, Guaza C, Borrell J. Neurobehavioral and immunological consequences of prenatal immune activation in rats. Influence of antipsychotics. Neuropsychopharmacology. 2007 Aug;32(8):1791-804. doi: 10.1038/sj.npp.1301292. Epub 2006 Dec 20. PMID 17180123
- [Background] Romero E, Guaza C, Castellano B, Borrell J. Ontogeny of sensorimotor gating and immune impairment induced by prenatal immune challenge in rats: implications for the etiopathology of schizophrenia. Mol Psychiatry. 2010 Apr;15(4):372-83. doi: 10.1038/mp.2008.44. Epub 2008 Apr 15. PMID 18414405
- [Background] Behrens MM, Ali SS, Dugan LL. Interleukin-6 mediates the increase in NADPH-oxidase in the ketamine model of schizophrenia. J Neurosci. 2008 Dec 17;28(51):13957-66. doi: 10.1523/JNEUROSCI.4457-08.2008. PMID 19091984

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Following a screening evaluation, participants will receive two infusions of Tocilizumab, one at baseline and another at week 4 of the study. All subjects will receive a 4 mg/kg infusion of Tocilizumab, the recommended starting dose for adults with rheumatoid arthritis.
  Tocilizumab: Therapeutic/Pharmacological Class of Drug:
  Tocilizumab is a recombinant humanized anti-human interleukin-6 (IL-6) receptor monoclonal antibody of the immunoglobulin (Ig) gamma-1 subclass.
  Type of Dosage Form:
  Concentrate for solution for infusion.
  Route of Administration:
  Intravenous (i.v.) infusion.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab: Following a screening evaluation, participants will receive two infusions of tocilizumab, one at baseline and another at week 4 of the study. All subjects will receive a 4 mg/kg infusion of tocilizumab, the recommended starting dose for adults with rheumatoid arthritis.
  Tocilizumab: Therapeutic/Pharmacologic Class of Drug:
  Tocilizumab is a recombinant humanized anti-human interleukin-6 (IL-6) receptor monoclonal antibody of the immunoglobulin (Ig) gamma-1 subclass.
  Type of Dosage Form:
  Concentrate for solution for infusion.
  Route of Administration:
  Intravenous (i.v.) infusion.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 35 [23 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) is the metric used to characterize cognition in this study. The BACS consists of 6 subscales: Verbal Memory (range 0-75), Working Memory (range 0-28), Motor Speed (range 0-100), Verbal Fluency (measure is total number of words generated in two 60 second trials), Attention and Processing speed (range 0-110), and Executive Function (range 0-22). For each subscale, higher scores reflect better cognition. For each subscale, a Standard Deviation Score was calculated based on normative data (Keefe et al. Norms and standardization of the Brief Assessment of Cognition in Schizophrenia (BACS). Schizophrenia Research 102 (2008) 108-115). The BACS composite score is calculated as the average Standard Deviation Score of the 6 subscale scores. The change in BACS composite score was calculated as the BACS composite score at 8 weeks minus the BACS composite score at baseline.
Time Frame: Change in BACS composite score from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Change in BACS Composite Score
Arm/Group | Tocilizumab
Number analyzed (Participants) | 6
Change in BACS Composite Score | 0.7 (0.4)

2. Secondary Outcome: Change in Total Psychotic Symptoms
Description: The Positive and Negative Symptoms Scale (PANSS) is the metric used to characterize psychotic symptoms in this study. The PANSS consists of 30 items, each scored 1-7. The range for the PANSS total score is 30-210. There are 3 subscales - PANSS positive score (range 7-49), PANSS negative score (range 7-49), and PANSS general score (range 16-112). PANSS total score is the summation of these 3 subscales. Higher values for the total and subscale scores reflect more severe psychopathology. A positive change in PANSS total score reflects an increase in psychopathology. A negative change in PANSS total score reflects a decrease in psychopathology.
Time Frame: Change in PANSS total score from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Change in PANSS Total Score
Arm/Group | Tocilizumab
Number analyzed (Participants) | 6
Change in PANSS Total Score | -2.6 (10.5)

ADVERSE EVENTS:
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=6)
Psychiatric Hospitalization (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No